CLINICAL TRIAL: NCT04711369
Title: Lasertherapy for Vulvodynia
Acronym: Lydia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 32-187 ex 19/20
Record Dates: First submitted 2020-12-15; First posted 2021-01-15 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Vulvodynia
Keywords: Erbium:Yag laser
MeSH Terms: conditions — Vulvodynia

STUDY DESIGN:
Intervention Model Description: Randomized double blinded sham-controlled clinical study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Sham-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (laser therapy) (Active Comparator): Participants allocated to the laser-therapy group will receive 2 laser treatments over a period of 3 months. Laser therapy will be performed according to a standardized protocol.
  Interventions: Device: Erbium:Yag laser
- Control group (sham laser therapy) (Sham Comparator): Participants allocated to the control group will receive 2 sham laser treatments over a period of 3 months. Laser therapy will be performed according to a standardized protocol.
  Interventions: Device: Sham Erbium:Yag laser

INTERVENTIONS:
Device: Erbium:Yag laser — Vulvovaginal laser therapies will be performed with the non-ablative 2940 nm Er:YAG laser (Smooth XS, Fotona, Slovenia) in the Renova mode according to the manufacturer's guidelines and recommendations. The spot size (diameter of the laser beam) is 7 mm, with a pulse at a frequency of 1.6 Hz, and a fluence (laser energy delivered per unit area) of 5.0 to 10.0 J/cm2.
  All sensitive/painful areas of the introitus will be treated, using 1-3 repetitions.
  In postmenopausal women with signs of atrophy, additional irradiation of the vaginal wall will be performed.
  Arms: Intervention group (laser therapy)
Device: Sham Erbium:Yag laser — Clinical examination and preparations will be identical to the intervention group. Sham laser treatments will be performed with the same laser and the same procedures. However, a specially devised placebo probe with a steel shutter, which blocks the emission of radiation, will be used. Women will therefore receive no therapeutic irradiation. Before treatment, a study assistant, who is aware of the study allocation, will prepare the laser with the placebo probe, which looks identically to the "normal" probe. The treating physician will not be aware of the study allocation and the type of probe in use.
  Arms: Control group (sham laser therapy)

SUMMARY:
The study aims to assess the efficacy, acceptance and safety profile of vulvovaginal laser therapy in women with vulvodynia.

DETAILED DESCRIPTION:
Randomized double blinded sham-controlled clinical study

Main hypothesis:

Laser therapy will be more effective than sham laser therapy in vulvar pain reduction measured by Q-tip test and tampon test

Secondary study hypotheses Laser therapy, in comparison to sham laser therapy

* will lead to more improvement of Sexual Health and HrQoL
* will have similar rates of side effects

ELIGIBILITY:
Inclusion Criteria:

* Women with vulvodynia (diagnosed according to the 2015 Consensus Terminology)
* multidisciplinary treatment for at least 3 months
* Informed consent

Exclusion Criteria:

* Current genital infection (i.e. candidiasis, herpes )
* Inflammatory vulvar disease/ dermatosis (i.e. lichen sclerosus, lichen planus)
* Neoplastic vulvar disease (e.g. HSIL Vulva, Paget disease)
* Recent vulvar trauma (i.e. bleeding, erosion or ulceration)
* Pudendal neuralgia
* Pregnancy, delivery <6 months
* Epilepsy or major neurologic or psychiatric morbidity
* Active systemic infection
* Previous treatment with ionizing radiation in the area to be treated
* History of wound healing disorders (i.e. hyperpigmentation, abnormal scarring)
* Fever
* Systemic or local autoimmune disorders
* History of photosensitivity disorder

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2021-01-15 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Change of Vestibular pain index | Baseline and final assessment (3 months).
  The Vestibular pain index is derived from the Q-tip test and the tampon test. A standardized Q-Tip test (MRC Systems GmbH, Heidelberg, Germany), developed for quantitative sensoric testing, will be used. Pain on six defined anatomical regions of the vulvar vestibule (at 2 ,5,6,7,10 and 12 o clock) will be assessed. Patients will be asked to rate the level of vulvar pain on a numeric rating scale (NRS) of 0 "none at all" to 10 "worst imaginable".
  The tampon test is a standardized tampon insertion and removal test.
  The vestibular pain index will be calculated as follows:
  (mean NRS score of the standardized Q-tip test (6 sites) + NRS score during the tampon test) / 2

SECONDARY OUTCOMES:
Change of pelvic floor muscle (PFM) function- PFM contraction strength | Baseline and final assessment (3 months).
  The Modified Oxford Scale (MOS) will be used to score maximal PFM contraction strength, ranging from 0 (no contraction) to 5 (strong contraction and lift).
Change of pelvic floor muscle (PFM) function- PFM tone | Baseline and final assessment (3 months).
  PFM tone will be scored on a 7-point PFM tone scale ranging from -3 (very hypotonic) to +3 (very hypertonic), with 0 representing a "normal" pelvic muscle tone.
Change of levator hiatal dimensions at rest | Baseline and final assessment (3 months).
  3D perineal ultrasound will be used to measure levator hiatal dimensions at rest
Change of levator hiatal dimensions at maximal voluntary contraction | Baseline and final assessment (3 months).
  3D perineal ultrasound will be used to measure levator hiatal dimensions at maximal voluntary contraction
Change of levator hiatal dimensions at maximal Valsalva maneuver | Baseline and final assessment (3 months).
  3D perineal ultrasound will be used to measure levator hiatal dimensions at maximal Valsalva maneuver
Change of Vaginal health score index (VHSI) | Baseline and final assessment (3 months).
  In postmenopausal women the VHSI will be performed to assess elasticity, fluid volume, pH, epithelial integrity and a moisture on a scale from 1 (none) to 5 (excellent) each. The sum score will be recorded.
Change of Sexual activity | Baseline and final assessment (3 months).
  Participants will be asked to complete a study diary and record whether they experienced sexual intercourse. Possible answers are: #1-"No, too painful" indicating that the woman could not accept an approach to physical intimacy because of pain, #2 -"No, not interested", indicating that the subject was not in the mood for sexual intimacy, #3-"No,no opportunity", indicating that her partner was not available, #4-"Yes" meaning that an attempt at sexual intercourse was made. If intercourse was attempted the level of pain during intercourse should be rated on a 0 - 10 NRS pain scale.
Change of Sexual Function | Baseline and final assessment (3 months).
  The German version of the Female Sexual Function Index (FSFI-d) will be used to assess women´s sexuality. The validated 19-item questionnaire examines several aspects of female sexuality, i.e. sexual arousal, orgasm and dyspareunia.
Change in Endometriosis Health Profile (EHP-30) | Baseline and final assessment (3 months).
  The EHP-30 consists of five scales -pain, control and powerlessness, emotional well-being, social support, and self-image (30 items) and a module with 23 items. The modular part consists of six scales - work, relationship with children, sexual intercourse, infertility, medical profession, and treatment.
Change in German Pain Assessment (assessed by Deutscher Schmerzfragebogen/DSF) | Baseline and final assessment (3 months).
  The DSF was developed for the comprehensive assessment and therapy planning of patients with chronic pain conditions. The modules on pain assessment (e.g. pain characteristics, relieving and aggravating factors) and on demographic information will be used.
Change in Patient Health Questionnaire (PHQ-D) | Baseline and final assessment (3 months).
  The PHQ-D is a sensitive screening tool for detecting depressive symptoms in a general patient population. The 9-item tool assesses the degree and severity of depression, and has been found to be a valid and useful tool for therapy evaluation
Change in Pain sensitivity questionnaire (PSQ) | Baseline and final assessment (3 months).
  The PSQ is an instrument for the assessment of pain sensitivity based on pain intensity self ratings of daily life situations
Change in Patient Global Impression of Improvement (PGI-I) | Baseline and final assessment (3 months).
  The Patient Global Impression of Improvement (PGI-I), a valid instrument with a 7-step Likert type response scale, will be used to assess subjective improvement after treatment. After three months, i.e. one month after the second laser therapy, women will be asked to rate the change in vulvar pain.
Change in Patient treatment satisfaction | Baseline and final assessment (3 months).
  Treatment satisfaction will be assessed using an adopted version of the "Fragebogen zur Patientenzufriedenheit - ZUF8". The questionnaire, the German version of the original "Client Satisfaction Questionnaire-CSQ8", is a tool for measuring global patient satisfaction at the end of inpatient treatment
Change in Treatment discomfort | Twice after treatment, one and two months after baseline
  At the end of each treatment session patients are asked to indicate the degree of discomfort during laser therapy on a NRS ranging from 0 "no discomfort" to 10 "worst possible discomfort"
Change in Treatment pain | Twice after treatment, one and two months after baseline
  At the end of each treatment session patients are asked to indicate the degree of pain during laser therapy on a NRS ranging from 0 "no pain" to 10 "worst possible pain".

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology/ Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No